CLINICAL TRIAL: NCT02005458
Title: Multi-center, Randomized, Open-labeled, Positive-controlled, Phase Ⅱ Study to Evaluate Efficacy and Safety of YPEG-rhG-CSF, Once-per-cycle, Comparing to PEG-rhG-CSF, Once-per-cycle, in Chemotherapy-induced Neutropenia of Patients With Malignancies Receiving Myelosuppressive Chemotherapy.
Brief Title: Safety and Efficacy of YPEG-rhG-CSF in Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1309CSF
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer; Breast Cancer
Keywords: Neutropenia; Febrile neutropenia; PEG-rhG-CSF; Myelosuppressive chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Neutropenia; Febrile Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- YPEG-rhG-CSF 20μg/kg (Experimental): 20μg/kg,single s.c. at 48hrs after chemotherapy for each experimental cycle
  Interventions: Drug: YPEG-rhG-CSF, 20μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
- YPEG-rhG-CSF 30μg/kg (Experimental): 30μg/kg,single s.c. at 48hrs after chemotherapy for each experimental cycle
  Interventions: Drug: YPEG-rhG-CSF, 30μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
- YPEG-rhG-CSF 45μg/kg (Experimental): 45μg/kg,single s.c. at 48hrs after chemotherapy for each experimental cycle
  Interventions: Drug: YPEG-rhG-CSF, 45μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
- PEG-rhG-CSF 100μg/kg (Active Comparator): 100μg/kg,single s.c. at 48hrs after chemotherapy for each experimental cycle
  Interventions: Drug: PEG-rhG-CSF, 100μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle

INTERVENTIONS:
Drug: YPEG-rhG-CSF, 20μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
  Arms: YPEG-rhG-CSF 20μg/kg
Drug: YPEG-rhG-CSF, 30μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
  Arms: YPEG-rhG-CSF 30μg/kg
Drug: YPEG-rhG-CSF, 45μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
  Arms: YPEG-rhG-CSF 45μg/kg
Drug: PEG-rhG-CSF, 100μg/kg, single s.c. at 48hrs after chemotherapy for each experimental cycle
  Arms: PEG-rhG-CSF 100μg/kg

SUMMARY:
This study is to examine which dose of YPEG-rhG-CSF, once-per-cycle, has similar efficacy and safety, comparing to PEG-rhG-CSF, once-per-cycle, in chemotherapy-induced neutropenia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small cell lung cancer or Breast cancer, and adequate for carboplatin combined with taxol or cyclophosphamide combined with pharmorubicin chemotherapy
* Karnofsky Score ≥ 70
* Life Expectancy > 3 months
* Age: 18～70yrs.
* Peripheral blood test: WBC≥3.5×106/mm3, PLT≥100×106/mm3, ANC≥1.5×106/mm3; Normal bone marrow function; Bone marrow biopsy shows active hematopoietic without cancer cells.
* Normal coagulation function, no evidences of hemorrhage tendency.
* No exiting diseases or condition that may influence drug absorption, distribution, metabolism, and excretion.
* Adequate liver, cardiac, kidney function. Indicators of liver function test ≤ 2.5ULN, Indicators of kidney function test ≤ 1ULN
* Understand and voluntarily sign an informed consent form.

Exclusion Criteria:

* Pregnant or lactating females
* Evidence of tumor metastasis in bone marrow
* Lack insight due to tumor metastasis in the central nervous system
* Prior bone marrow transplant or stem cell transplant
* Infective symptom before enrollment into this study
* Other malignancy history
* Known hypersensitivity to any component of the drug(e.g. rh-G-CSF) that to be administered
* Subject enrolled in any other investigational drug or device trial within 3 months of informed consent date
* Drug abuser or alcoholist
* Prior radiotherapy or expected to received radiotherapy
* Unstable or uncontrolled cardiac or hypertension
* Other conditions which in the opinion of the investigator preclude enrollment into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Grade 3 &4 neutropenia, and median duration of neutropenia in the two experimental cycles | 21 day
  Grade 3 and 4 neutropenia means absolute neutrophil count is less than 1000/mm3 and 500/mm3 , respectively

SECONDARY OUTCOMES:
Incidence of febrile neutropenia in the two experimental cycles | 21 day
  Febrile neutropenia means absolute neutrophil count is less than 500/mm3 or absolute neutrophil count between 500/mm3 and 1000mm3 but probably to decline to less than 500mm3 within 48hrs, and body temperature is higher than 38.5 degrees celsius or higher than 38.0 degrees celsius and lasting for more than 1hr
Diversification of neutrophil in the two experimental cycles | 21 day

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (12):
- China (12):
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Shaaxi Provincial Tumor Hospital, Xi'an, Shaanxi
  - Cancer Institute and Hospital, CAMS, Beijing
  - Fujian cancer hospital, Fuzhou
  - Fujian Medical University Union Hospital, Fuzhou
  - Fuzhou General Hospital of Nanjing Military Command, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Shanghai Changzheng Hospital, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Tongji Hospital, Tongji Medical College Huazhou University of Science & Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Zhejiang cancer hospital, Zhejiang